CLINICAL TRIAL: NCT02012023
Title: Use of One Kind of Controllable Tube Ileostomy to Protect Anastomotic Leakage in the Low Rectal Cancer.
Brief Title: Use of One Kind of Controllable Tube Ileostomy in the Low Rectal Cancer
Acronym: CTI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Hua hanju, Doctor, First Affiliated Hospital of Zhejiang University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Controllable tube ileostomy
Record Dates: First submitted 2013-12-04; First posted 2013-12-16 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-07

CONDITIONS: Rectal Neoplasms; Low Anterior Resection
Keywords: Low anterior resection; Anastomotic leakage; Defunctioning stoma; Controllable tube ileostomy; Loop ileostomy
MeSH Terms: conditions — Rectal Neoplasms; Anastomotic Leak | interventions — Ileostomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Controllable tube ileostomy (Experimental): After LAR, the experimental group accepted controllable tube ileostomy.
  Interventions: Device: Low anterior resection; Device: tube ileostomy; Device: remove the tube ileostomy
- Loop ileostomy (Active Comparator): After LAR, the experimental group accepted loop ileostomy.
  Interventions: Device: Low anterior resection; Device: loop ileostomy; Device: accept reversal operation

INTERVENTIONS:
Device: Low anterior resection
Device: tube ileostomy
  Arms: Controllable tube ileostomy
Device: loop ileostomy
  Arms: Loop ileostomy
Device: accept reversal operation
  Arms: Loop ileostomy
Device: remove the tube ileostomy
  Arms: Controllable tube ileostomy

SUMMARY:
Most surgeons suggest the use of fecal diverting to address the high morbidity and mortality associated with anastomotic leakage (AL) in patients with high risk factors on AL who are undergoing low anterior resections(LAR). This exploratory study was conducted to evaluate the efficacy and safety of one kind of controllable tube ileostomy(CTI), which was designed to protect rectal anastomosis in patients with high risk factors on AL. Results of SCCI were compared to those of the loop ileostomy (LI) method.

In fact when we told the patients about the tube ileustomy's effect and risk, almost all the almost all of my patients like to choose tube ileustomy(I have study this method for long time and have good expeience, and my patients either choose tube ileostomy directly or let me do the choice.) So I gave all the patients who meet the requirenments all tube ileustomy and have no control group.

DETAILED DESCRIPTION:
After low anterior resection(LAR), a double row of concentric purse-string sutures were placed in the ileum wall using 3-0 absorbable suture. The diameters of the purse-string rings were about 10 mm and 20 mm, respectively. The investigators then made a small incision within the inner purse-string and inserted the trachea cannula into the proximal end of the ileum. The inner purse-string suture then was tied, followed by the outer purse-string suture. The outer purse string should capsulate the inner purse string to prevent leakage. Normal saline was injected into the air bag until the ileum wall. The investigators will test the pressure of airbag, and control the pressure of airbag from 30-40cmHg. The investigators then pulled the cannula out through the abdominal wall. The incision site in the ileum was approximated to the inner abdominal wall and extraperitonized by fixing the mobilized ileum wall around the cannula to the inner abdominal wall. This was accomplished using 3-4 interrupted sutures.

In the CTI group, the tube will be removed after 3-4 weeks. If anastomotic leakage occurred, the investigators will test the airbag pressure and keep the pressure during 30-40cmHg. Because with time went on, the ileum will dilated , the airbag pressure will go down, then the feces may go through the airbag plane and flow into colon and the tube ileostomy will lose its defunctioning effect.When the investigators control the airbag pressure, we can control the defunctioning effect of tube stomy. So it is called controllable tube ileostomy. The investigators will keep the tube until the anastomotic leakage was cured.

ELIGIBILITY:
Inclusion Criteria:

* Rectal Tumor After Low Anterior Resection the Anastomosis Located extraperitoneal
* Patients Agreed to Undergo the tube ileostomy or loop ileostomy Procedure

Exclusion Criteria:

* Bowel Preparation is not Satisfied Before Operation
* Blood lose is more than 1500ml during operation
* Critical incident during operation
* The vagina or bladder is seriously damaged and the fix is not satisfied.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-01; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
anastomotic leakage | about in 3 months after operaion
  Anastomotic leakage(AL) is the main complication after LAR.AL is defined as a defect of intestinal wall integrity at the colorectal or coloanal anastomotic site (including suture and staple lines of the neorectal reservoirs) leading to communication between intra- and extraluminal compartments.
reoperation rate | about 3 months after operation
  When AL occurred, whether this patient need reoperation is determined by the clinical manifestation. Reoperation rate and mortality are two key index to evaluate the effect and safety of cannula ileostomy.
mortality | about 3 months after operation

SECONDARY OUTCOMES:
ileus rate | during the follow time(about 6 months after operaion)
  Another main operation complication was intestinal obstruction. Ileus conclude two types: temporally ileus and intractable ileus. Temporally ileus can be treated by conservative treatment and intractable ileus need reoperation.Ileus usually is caused by intestinal adhesion. But in CTI group, ileus maybe caused by the cannula obstruction.
operation data | durting the operation time (about 1-5 h)
  including operation method, time, blood loss et al.

OTHER OUTCOMES:
hospital stays | from admission time to discharge time(about 7-14days)
  In loop ileostomy group, hospital stays and costs include the readmission to close the stoma.
hospital costs | from admission time to discharge time(about 7-14days)
  In loop ileostomy group, hospital stays and costs include the readmission to close the stoma.

CONTACTS AND LOCATIONS:
Overall Officials: Hua Hanju, Doctor, Principal Investigator — Zhejiang University
Locations (1):
- Department of Colorectal Surgery, First Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes